CLINICAL TRIAL: NCT01272895
Title: Evaluation of Endothelial Progenitor Cell (EPC) Capturing (GENOUS) Stent After Coronary Stenting Utilizing Optical Coherence Tomography (OCT): the EGO Study
Brief Title: OCT Evaluation of Early Healing of EPC Capturing (GENOUS) Stent (EGO Study)
Acronym: EGO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Stephen Lee (Other)
Responsible Party: Sponsor-Investigator, Prof. Stephen Lee, Professor and Chief, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 10-256 (IRB HKU)
Record Dates: First submitted 2010-12-28; First posted 2011-01-10 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Artery Disease
Keywords: OCT images; Stent strut coverage; Endothelialization; Neointimal thickness, area and hyperplasia; Stent malapposition
MeSH Terms: conditions — Coronary Artery Disease; Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GENOUS stent (Experimental)
  Interventions: Device: Coronary Intervention (GENOUS stent)

INTERVENTIONS:
Device: Coronary Intervention (GENOUS stent) — GENOUS stent (Coronary Intervention)
  Other Names: EPC capturing Genous R-Stent

SUMMARY:
All patients who have received GENOUS stent implantation at Queen Mary Hospital for treatment of ischemic heart disease are eligible for this study. Those with clinical indications to undergo restudy coronary angiogram or staged procedure PCI will be primarily recruited into this study.

Optical coherence tomography (OCT) will be performed early after stent implantation to evaluate vascular healing response and neointimal coverage.

DETAILED DESCRIPTION:
The GENOUS Stent is a bio-engineered 316L stainless steel coronary stent with a biocompatible circumferential coating of anti-CD34 antibody, and will bind to and therefore capture the circulatory endothelial progenitor cells (EPC) which have CD34 antigen on the surface. Immobilization of EPCs on the stent surface will encourage differentiation and proliferation of the EPCs into endothelial and neointimal layer. This stent has been used extensively in 180 patients at Queen Mary Hospital with critical coronary stenosis.

Animal model has demonstrated that a functional endothelial layer could be formed as soon as 24 to 48 hours after GENOUS stent implantation (1). The HEALING-FIM registry has shown that GENOUS stent is clinically safe and effective in the treatment of coronary stenosis (2). Recent reports have further confirmed its efficacy in patients with acute coronary syndrome requiring urgent revascularization (3,4).

Intracoronary frequency domain optical coherence tomography (FD-OCT) is a simple catheter-based imaging technique using optic fibre to achieve very detailed assessment (resolution down to 10 microns) of the stents, in terms of stent apposition, early neointimal coverage (enhanced endothelialization) and late stent neointimal growth (restenosis). It is performed as part of the routine cardiac catheterization procedure and provides high-resolution cross sectional images of the coronary arteries. OCT has been shown to be safe in clinical practice (5). The LightLab C7XR OCT System (Frequency Domain OCT) is a commercially available product with CE Mark and FDA approval, and is being used in our EGO Study. The Dragonfly OCT catheter used is a non-occlusive optic fibre which is extremely small and flexible, and will pose absolutely no additional risk to the patient under treatment, other than those inherent risks of a standard angioplasty procedure.

Despite data in animal model showed a fast and complete endothelization, there is no study to verify and investigate on such healing benefits in human patients. Therefore, if endothelization and early neointimal healing benefits of the GENOUS stent can be evaluated by a reliable imaging technique, further studies can be carried out to extend the benefits of the EPC capturing capacity.

ELIGIBILITY:
Inclusion Criteria:-

1. Patients aged 18-85 years old who received GENOUS stent treatment for ischemic coronary disease, and
2. Clinically indicated for a follow-up coronary angiogram or repeated (staged) coronary interventions within 3 months.

Exclusion Criteria:-

Patients who refuse to consent to coronary angiogram or coronary angioplasty.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Percentage stent coverage by OCT in early phases. | At 2nd, 3rd, 4th, 5th, and 6th weeks after stent implantation
  Percentage stent strut coverage at weekly intervals from 2nd to 6th week after EPC capturing stent implantation as assessed by OCT according to our OCT Early Coverage Classification.

SECONDARY OUTCOMES:
Other OCT Findings | At 2nd, 3rd, 4th, 5th, and 6th week
  Neointimal thickness, neointimal area, late lumen loss, and percentage strut malapposition at the time of OCT follow up observed between the 5 different weekly groups.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen WL Lee, MD FRCP FACC, Principal Investigator — Queen Mary Hospital, The University of Hong Kong
Locations (1):
- Division of Cardiology, Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Result] Aoki J, Serruys PW, van Beusekom H, Ong AT, McFadden EP, Sianos G, van der Giessen WJ, Regar E, de Feyter PJ, Davis HR, Rowland S, Kutryk MJ. Endothelial progenitor cell capture by stents coated with antibody against CD34: the HEALING-FIM (Healthy Endothelial Accelerated Lining Inhibits Neointimal Growth-First In Man) Registry. J Am Coll Cardiol. 2005 May 17;45(10):1574-9. doi: 10.1016/j.jacc.2005.01.048. PMID 15893169
- [Result] Co M, Tay E, Lee CH, Poh KK, Low A, Lim J, Lim IH, Lim YT, Tan HC. Use of endothelial progenitor cell capture stent (Genous Bio-Engineered R Stent) during primary percutaneous coronary intervention in acute myocardial infarction: intermediate- to long-term clinical follow-up. Am Heart J. 2008 Jan;155(1):128-32. doi: 10.1016/j.ahj.2007.08.031. Epub 2007 Nov 26. PMID 18082503
- [Result] Miglionico M, Patti G, D'Ambrosio A, Di Sciascio G. Percutaneous coronary intervention utilizing a new endothelial progenitor cells antibody-coated stent: a prospective single-center registry in high-risk patients. Catheter Cardiovasc Interv. 2008 Apr 1;71(5):600-4. doi: 10.1002/ccd.21437. PMID 18360849
- [Result] Yamaguchi T, Terashima M, Akasaka T, Hayashi T, Mizuno K, Muramatsu T, Nakamura M, Nakamura S, Saito S, Takano M, Takayama T, Yoshikawa J, Suzuki T. Safety and feasibility of an intravascular optical coherence tomography image wire system in the clinical setting. Am J Cardiol. 2008 Mar 1;101(5):562-7. doi: 10.1016/j.amjcard.2007.09.116. Epub 2008 Jan 10. PMID 18307999
- [Result] Prati F, Cera M, Ramazzotti V, Imola F, Giudice R, Albertucci M. Safety and feasibility of a new non-occlusive technique for facilitated intracoronary optical coherence tomography (OCT) acquisition in various clinical and anatomical scenarios. EuroIntervention. 2007 Nov;3(3):365-70. doi: 10.4244/eijv3i3a66. PMID 19737719